CLINICAL TRIAL: NCT04899531
Title: Longitudinal PANGeA Mass Measurement - Physical Activity and Nutrition for Quality Ageing
Brief Title: PANGeA - Physical Activity and Nutrition for Quality Ageing
Acronym: PANGeA_MM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Science and Research Centre Koper (Other)
Responsible Party: Principal Investigator, Rado Pisot, Professor, Science and Research Centre Koper
Other Study IDs: PANGeA MM
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Aging; Sarcopenia; Cognitive Decline
Keywords: elderly; longitudinal; physical activity; cognition; dietary habits
MeSH Terms: conditions — Sarcopenia; Cognitive Dysfunction; Motor Activity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Longitudinal observation: No specific intervention, pre-post measurements only
  Interventions: Other: Longitudinal observation

INTERVENTIONS:
Other: Longitudinal observation — No specific intervention, longitudinal (pre-post measurements) only

SUMMARY:
General objectives of the project

Defining healthy ageing factors; Setting up content-related bases of the international excellence centre (SLO-ITA) in the field of health of elderly citizens; Raising awareness on the significance of healthy ageing, social inclusion and mobility of less privileged populations (the elderly); Reducing the costs of health care; Connecting the existing health care, social and private entities and improving their mutual coordination.

DETAILED DESCRIPTION:
Physical activity, dietary habits, social and private entities strongly affect the quality of health and quality of life of the elderly. The main object of this study will be to evaluate physical and cognitive performance in combination with physical activity and dietary habits of the elderly. The investigators are interested in longitudinal monitoring of the elderly that participated in measurements in 2013 and measurements after a decade. The results of this study will give important epidemiological information about physical and cognitive status, health status in combination with physical activity which occurs in a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* singed written consent
* age above 60
* healthy

Exclusion Criteria:

* severe musculoskeletal injuries
* inability to follow instructions when performing the test

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All males and females who participated in PANGeA mass measurements in 2013 will bi considered in the study.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2013-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Grip strength | change in grip strength between two observational time points (pre-post 8-10years)
  Grip strength measured using a hand-held dynamometer

SECONDARY OUTCOMES:
Gait speed | change in gait speed between two observational time points (pre-post 8-10years)
  Gait speed measured for four meters self selected speed

CONTACTS AND LOCATIONS:
Overall Officials: Rado Pišot, PhD, Study Director — Science and Research Centre Koper
Locations (1):
- Science and research centre Koper, Koper, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Teraz K, Marusic U, Kalc M, Simunic B, Pori P, Grassi B, Lazzer S, Narici MV, Blenkus MG, di Prampero PE, Reggiani C, Passaro A, Biolo G, Gasparini M, Pisot R. Sarcopenia parameters in active older adults - an eight-year longitudinal study. BMC Public Health. 2023 May 19;23(1):917. doi: 10.1186/s12889-023-15734-4. PMID 37208654